CLINICAL TRIAL: NCT03043079
Title: Ultrasound Assessment of Ventral Hernia Defects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, John Fischer, MD, MPH, Assisstant Professor of Surgery, University of Pennsylvania
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 823896
Record Dates: First submitted 2017-01-24; First posted 2017-02-03 (Estimated); Results first posted 2020-03-24 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Ventral Incisional Hernia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Ventral Hernia (Experimental): Twenty-five patients diagnosed with ventral hernia
  Interventions: Diagnostic Test: Ultrasound Acoustic Radiation Forced Impulse Shear Wave Velocity
- Healthy Volunteers (Other): Twenty-five volunteers without ventral hernia
  Interventions: Diagnostic Test: Ultrasound Acoustic Radiation Forced Impulse Shear Wave Velocity
- Active Health Volunteers (Other): Ten healthy volunteers with an International Physical Activity Questionnaire (IPAQ) with the scoring result of High or Vigorous Intensity
  Interventions: Diagnostic Test: Ultrasound Acoustic Radiation Forced Impulse Shear Wave Velocity

INTERVENTIONS:
Diagnostic Test: Ultrasound Acoustic Radiation Forced Impulse Shear Wave Velocity — Abdominal Ultrasound Acoustic Radiation Forced Impulse Shear Wave Velocity (ARFI-SWV)

SUMMARY:
Quantitative radiographic imaging holds promise as a novel and innovative strategy to assess ventral hernia patients. Assessing abdominal wall changes surrounding ventral hernia using shear wave velocity values measured with ultrasound will identify features of the abdominal wall that differ between healthy volunteers and subjects scheduled to have ventral hernia repair. Through the use of ultrasound including shear wave velocity measurements, the abdominal wall of 25 subjects scheduled to have ventral hernia repair will be compared to those of 35 healthy volunteers. The ultrasound measurements will elucidate if ventral hernia affects abdominal wall elasticity and effect surgical outcomes.

DETAILED DESCRIPTION:
ARFI-SWV Ultrasound holds promise as an inexpensive, noninvasive, point-of-care diagnostic tool for pre-operatively predicting successful hernia repair. The investigators propose to develop and refine a quantitative ultrasound protocol to measure abdominal wall features suitable for predicting successful closure of the midline fascia. ARFI-SWV ultrasound represents a novel and intriguing modality for real time visualization and characterization of changes in the biomechanical properties of diseased musculoskeletal tissues.

In this study, ARFI-SWV ultrasound is hypothesized to preoperatively measure the stiffness in the lateral abdominal wall as an estimation for mobility during hernia repair. Preoperatively evaluating hernia severity through ARFI-SWV ultrasound will be performed to identify mechanical characteristics of the abdominal musculature to predict success of midline fascial re-approximation in hernia patients. The study proposes to compare ultrasound images and associated shear wave velocity measurements between 35 healthy volunteers and 25 subjects undergoing surgical repair for ventral hernia. Subjects with ventral hernia will undergo imaging no earlier than two weeks prior to elective hernia repair and again postoperatively within six months following repair at a standard followup visit. Statistical analysis will determine if there is a significant difference in the abdominal wall stiffness, represented by the ultrasound shear wave velocity measurements, between the healthy subjects and the subjects with ventral hernia. Further analysis will determine if there is any statistically significant relationship between abdominal wall stiffness of subjects with ventral hernia and surgical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* male or female between 20-70 years of age
* healthy volunteer or seeking elective ventral hernia repair

Exclusion Criteria:

* pregnant women

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-09-15 (Actual); Study Completion 2017-09-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania Health System, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data to outside researchers at the end of the study. Any data shared will be de-identified.

RESULTS

PARTICIPANT FLOW:
Groups:
- Ventral Hernia: Twenty-One patients diagnosed with ventral hernia
  Ultrasound Acoustic Radiation Forced Impulse Shear Wave Velocity: Abdominal Ultrasound Acoustic Radiation Forced Impulse Shear Wave Velocity (ARFI-SWV)
- Healthy Volunteers: Fourteen volunteers without ventral hernia
  Ultrasound Acoustic Radiation Forced Impulse Shear Wave Velocity: Abdominal Ultrasound Acoustic Radiation Forced Impulse Shear Wave Velocity (ARFI-SWV)
Period: Overall Study
Arm/Group | Ventral Hernia | Healthy Volunteers | Active Health Volunteers
Started (We originally wanted 25 healthy/active volunteers. We divided that up into 15 healthy and 10 active.) | 21 | 14 | 10
Completed | 21 | 14 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Demographic data and shear wave velocity measurements were taken from each subject
Groups:
- Total: Total of all reporting groups
Arm/Group | Ventral Hernia | Healthy Volunteers | Active Health Volunteers | Total
Number analyzed (Participants) | 21 | 14 | 10 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 16 | 12 | 10 | 38
  >=65 years | 5 | 2 | 0 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.3 (7.9) | 60.5 (5.4) | 27.0 (3.17) | 48.6 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 8 | 4 | 23
  Male | 10 | 6 | 6 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 5 | 4 | 0 | 9
  White | 16 | 9 | 7 | 32
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 21 | 14 | 10 | 45
9L4 No Pressure External Oblique Shear Wave Velocity [Mean (Full Range); unit: meters per second] — For this measurement, a 9L4 probe is applied to the subjects abdomen without any pressure from the examiner, while the subject is holding end expiration. The shear wave velocity (m/s) is measured along the subject's external oblique muscle.
  meters per second | 1.94 [1.3 to 2.8] | 1.9 [1.2 to 2.83] | 1.97 [1.44 to 2.89] | 1.9 [1.08 to 2.89]

OUTCOME MEASURES:

1. Primary Outcome: Difference in the Shear Wave Velocity Measurements in the Abdominal Wall Between Ventral Hernia and Healthy Abdominal Wall
Description: Differences in the shear wave velocity measurements in the abdominal wall of healthy and ventral hernia patients
Time Frame: study intiation ultrasound scan lasting up to 45 minutes
Population: 21 ventral hernia age and BMI matched to 14 health volunteers with 10 active volunteers
Measure: Mean (Standard Deviation); unit: meters per second
Arm/Group | Ventral Hernia | Healthy Volunteers | Active Health Volunteers
Number analyzed (Participants) | 21 | 14 | 10
meters per second | 1.89 (.31) | 1.92 (.46) | 1.89 (.13)

2. Secondary Outcome: Difference in Shear Wave Velocity Measurement in the Abdominal Wall Pre and Post Hernia Repair
Description: Differences in the shear wave velocity measurements in the abdominal wall of preoperative hernia scan and postoperative scan 26 weeks after surgical ventral hernia repair
Time Frame: through study completion, an up to 26 weeks postoperative
Measure: Mean (Standard Deviation); unit: meters per second
Arm/Group | Ventral Hernia
Number analyzed (Participants) | 21
meters per second | 1.726 (0.36)

3. Secondary Outcome: Incidental Findings and Ultrasound Safety
Description: Any reported incidental findings or health related issues from being subjected to the study-related ultrasound imaging
Time Frame: 1 year
Measure: Number; unit: Participants
Groups:
- Ventral Hernia: Twenty-one patients diagnosed with ventral hernia
  Ultrasound Acoustic Radiation Forced Impulse Shear Wave Velocity: Abdominal Ultrasound Acoustic Radiation Forced Impulse Shear Wave Velocity (ARFI-SWV)
  No adverse events Related to study. No incidental findings from the Ultrasound
Arm/Group | Ventral Hernia
Number analyzed (Participants) | 21
Participants | 0

ADVERSE EVENTS:
Time Frame: Hernia patients were followed for adverse events for an average of 12 months. There were seen in the outpatuent clinic following typical standard of care guidelines, which is typically 2 weeks and 3 months. Healthy and active volunteers were followed during the initial ultrasound, up to 45 minutes.
Description: Adverse events were defined as any event that harmed subjects related to the study protocol. Adverse events related to the hernia surgery itself were not included in the study adverse events as the surgery plan was not affected by study participation. All subjects got the same surgical care that they would have if they were not enrolled in the study.
Groups:
- Ventral Hernia: Twenty-one patients diagnosed with ventral hernia
  Ultrasound Acoustic Radiation Forced Impulse Shear Wave Velocity: Abdominal Ultrasound Acoustic Radiation Forced Impulse Shear Wave Velocity (ARFI-SWV)
  No adverse events Related to study
- Healthy Volunteers: Fourteen volunteers without ventral hernia
  Ultrasound Acoustic Radiation Forced Impulse Shear Wave Velocity: Abdominal Ultrasound Acoustic Radiation Forced Impulse Shear Wave Velocity (ARFI-SWV)
  No adverse events Related to study
- Active Health Volunteers: Ten healthy volunteers with an International Physical Activity Questionnaire (IPAQ) with the scoring result of High or Vigorous Intensity
  Ultrasound Acoustic Radiation Forced Impulse Shear Wave Velocity: Abdominal Ultrasound Acoustic Radiation Forced Impulse Shear Wave Velocity (ARFI-SWV)
  No adverse events Related to study
Arm/Group | Ventral Hernia | Healthy Volunteers | Active Health Volunteers
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/14 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/14 | 0/10
Other Adverse Events (participants affected / at risk) | 0/24 | 0/14 | 0/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ventral Hernia (N=24) | Healthy Volunteers (N=14) | Active Health Volunteers (N=10)
Incidental Finding (Investigations) | 0 (0) | 0 (0) | 0 (0) — Any incidental findings that noted during study related ultrasound and required further clinical workup

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-12-09): https://cdn.clinicaltrials.gov/large-docs/79/NCT03043079/Prot_SAP_000.pdf